CLINICAL TRIAL: NCT03664245
Title: DetermInants of Antimicrobial Use aNd De-escalAtion in Critical Care (DIANA Study)
Brief Title: DetermInants of Antimicrobial Use aNd De-escalAtion in Critical Care
Acronym: DIANA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-20
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: Critically ill patients receiving empirical antibiotic therapy for suspected or confirmed infections at the Intensive Care Unit

SUMMARY:
Appropriate initial antibiotic therapy is crucial in the treatment of severe infections in patients with intensive care. Adequate spectrum and appropriate doses are the keys to achieving the therapeutic goal. Despite broad consensus on the spectrum and timing of antimicrobial therapy, antibiotic use varies according to various parameters including choice, dose, method of administration, duration of antibiotic therapy and de-escalation. an empirical attitude.

Therapeutic de-escalation is considered essential for the use of antibiotics and is now clearly established by different consensus. However, routine de-escalation has recently been questioned in a randomized, controlled study that did not demonstrate non-inferiority of de-escalation with an increase in the number of days of antibiotic therapy associated with an increased number of days. superinfection.

The components of the de-escalation described in the literature, are based on the reduction of the number of antibiotics, the strict observance of the spectrum of the antibiotic, the reduction of use of the antibiotic, the stopping of any inappropriate antibiotic treatment ( lack of in vitro activity).

De-escalation can be considered in different ways; there are significant variations between hospitals, countries, teams. A large European multicenter cohort is needed.

The main objective of this study is to describe empiric antibiotic therapy in intensive care and the modalities of de-escalation.

DETAILED DESCRIPTION:
Appropriate initial antibiotic therapy is crucial in the treatment of severe infections in patients with intensive care. Adequate spectrum and appropriate doses are the keys to achieving the therapeutic goal. Despite broad consensus on the spectrum and timing of antimicrobial therapy, antibiotic use varies according to various parameters including choice, dose, method of administration, duration of antibiotic therapy and de-escalation. an empirical attitude.

Therapeutic de-escalation is considered essential for the use of antibiotics and is now clearly established by different consensus. However, routine de-escalation has recently been questioned in a randomized, controlled study that did not demonstrate non-inferiority of de-escalation with an increase in the number of days of antibiotic therapy associated with an increased number of days. superinfection.

The components of the de-escalation described in the literature, are based on the reduction of the number of antibiotics, the strict observance of the spectrum of the antibiotic, the reduction of use of the antibiotic, the stopping of any inappropriate antibiotic treatment ( lack of in vitro activity).

De-escalation can be considered in different ways; there are significant variations between hospitals, countries, teams. A large European multicenter cohort is needed.

The main objective of this study is to describe empiric antibiotic therapy in intensive care and the modalities of de-escalation (rate of de-escalation, incidence of mortality, length of stay in intensive care unit, relapse, rate of superinfection)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patient is admitted to an ICU and has an anticipated need of ICU support of at least 48 hours.
* Patient has a suspected or confirmed bacterial infection (community-, healthcare-, hospital- or ICU-acquired).
* Empirical antibiotic therapy is started for this infection at any time in the ICU or no more than 24 hours prior to ICU admission. If the initial antibiotic therapy is considered inadequate and another empirical scheme is chosen at ICU admission, this will be the empirical antibiotic of the study.
* Causative pathogen and susceptibility are unidentified at time of initiation of the antibiotic therapy.

Exclusion Criteria:

* Previous inclusion in this study for another infection - each patient can only be included once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients receiving empirical antibiotic therapy for suspected or confirmed infections at the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Antibiotic used | 28 days
  analyse the list of antibiotics used during 28 days

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, MD, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France